CLINICAL TRIAL: NCT05388734
Title: Shared Decision Making on Care Pathways and CAMs: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other); Laboratoire TIMC-IMAG (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A03027-34
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Non-metastatic; Newly Diagnosed; Feasibility Study
Keywords: Complementary and Alternative Medicine (CAM); breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, before-and-after, comparative, prospective, single-center, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before group (No Intervention): Patients in the before group are recruited during the first 4 months of the study and will not benefit from the alternative medicine education consultation
- After Group (Active Comparator): Patients in the front group are recruited from the 5th month of the study and will benefit from the alternative medicine education consultation
  Interventions: Other: alternative medicine education consultation

INTERVENTIONS:
Other: alternative medicine education consultation — The intervention will consist in a 1h30 individual consultation with a GP physician. Patients will be able to ask any questions they have regarding treatments for their breast cancer delivered outside of the hospital. Topics such as benefit-risk ratios, placebo effects and expectancies from CAM will be discussed with the patients. This consultation will promote a shared-decision model to help patients better discuss these matters with their healthcare providers.
  Arms: After Group

SUMMARY:
Shared Decision Making on Care Pathways and alternative and complementary medicine (CAMs) : A Pilot Study.

Study whose aim is to evaluate the feasibility of a study proposing a therapeutic education consultation leaning on the usual care pathway by estimating the recruitment capacity over 4 months as well as the acceptance rate of the study among patients diagnosed with breast cancer.

DETAILED DESCRIPTION:
The use of alternative and complementary medicine (CAMs) has been steadily increasing for several years. Certain populations are more likely than others to use this type of care, including breast cancer patients, for whom the rate of use is close to 90%. However, these populations are those for whom the risks associated with this type of care are the highest. In addition, patients rarely discuss alternative and complementary medicine (CAMs) with conventional care teams. As a result, patients often place unreasonable expectations on alternative and complementary medicine (CAMs) and at the same time put themselves in risky situations.

The aim of this project is to help breast cancer patients better orient themselves in their care pathway and in particular with regard to the plethora of alternative and complementary medicine (CAMs) available. They could therefore make an informed decision to seek (or not) treatment. In order to reach a shared decision, a consultation will be offered to patients with the objective of discussing their past recourse, their knowledge of the care pathway, their fears and their aspirations with regard to alternative and complementary medicine (CAM). Epistemological concepts (self-efficacy, placebo, benefit-risk ratio, etc.) will be discussed in order to allow these elements to be transposed throughout their care.

The impact of this consultation on compliance with conventional treatment, satisfaction with the treatment as a whole and communication with the rest of the health care team will be evaluated. A before/after methodology will first allow us to evaluate the values taken by our judgement criteria in the usual care pathway and then in the innovative care pathway proposed by the intervention. This study will allow us to establish the feasibility of a future research project of larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients recently diagnosed with breast cancer at Grenoble Alpes University Hospital
* In situ or invasive breast cancer, locally advanced but without metastasis, demonstrated on histology
* ECOG ( Eastern Cooperative Oncology Group) performance status 0, 1 or 2
* Cancer treated with chemotherapy, radiotherapy and/or surgery
* Having signed an informed consent after information, being of age and able to express consent, affiliated to a social security system

Exclusion Criteria:

* Pregnant, breastfeeding or parturient women
* women who do not speak French;
* patients participating in another research protocol
* Metastatic breast cancer, diagnosed psychiatric pathologies that make it impossible to perform the procedure, history of cancer except for cervical cancer in situ or basal cell cancer
* Subjects in a period of exclusion from another study,
* Subject under administrative or judicial supervision
* Subject unable to be contacted in case of emergency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a study proposing a therapeutic education consultation linked to the usual course of care | 8 month
  The investigators wish know the recruitment capacity in this study. To do this, the investigators will estimate the number of people included over 8 months (time of recruitment in the study).

SECONDARY OUTCOMES:
Evaluate literacy in the care pathway. | inclusion, 6 month
  "Health Literacy Questionnaire" (HLQ) at 6 month post intervention. Questionnaire contains 2 parts : P1 with 23 questions, and P2 with 21 questions.
  Coding:
  P1Q1 to P1Q23
  * Strongly Disagree = 1
  * Disagree = 2
  * Agree = 3
  * Strongly Agree = 4
  P2Q1 to P2Q21
  * Cannot do or always difficult, = 1
  * Usually difficult = 2
  * Sometimes difficult = 3
  * Usually easy = 4
  * Always easy = 5
  The HLQ consists of 9 scales representing 9 dimensions of health literacy. Each HLQ scale has 4-6 items. The HLQ does not provide one overall summative score. The scoring of the HLQ is 9 scale scores, calculated by averaging the item scores within each scale with equal weighting. The 9 scale scores will reflect a person's strengths and needs in the different dimensions of health literacy.
  For Scales 1 to 5, the score range is between 1 and 4 For Scales 6 to 9, the score range is between 1 and 5
Satisfaction with improvement in orientation to the care pathway | 6 month
  To assess the HQL (Health Literacy Questionnaire) Minimal Clinically Interesting Difference at 6 months after the intervention.
  The investigators wish to assess the Minimal Clinically Interesting Difference at 6 months after the intervention by comparing the response about the satisfaction with improvement in orientation to the care pathway (0: No improvement, 1 : Slight improvement, 2 : Good improvement, 3 : Excellent improvement) " to the HLQ dimensions of interest.
Success in orienting to the care pathway | inclusion, 6 month
  The investigators wish to assess PALS by comparing the response to the question "Do you feel able to learn about services and supports to ensure that all your health needs are met? ( YES/NO)" to the HLQ dimensions of interest.
  PALS will be binary, either patients feel able to orient themselves in the care pathway or they do not feel able to do so
Assess satisfaction with the current care pathway | 6 month
  Bilateral 6-item Likert scale at 6 months after surgery (-3: very dissatisfied to +3 very satisfied )
Collect the patient experience | 6 month
  Semi-directive interview conducted at 6 months after the intervention. This interview will be carried out only for some patients of the study until data saturation.
To assess patient adherence, patient believes in the mechanics of TACs operation. | inclusion, 6 month
  CHBQ questionnaire completed at inclusion (pre-intervention) and at 6 months (post-intervention by the patient.
  This questionnaire is composed of 10 propositions. The total score varies between 10 (total disagreement with all the proposals) and 70 (total agreement with all the proposals). The authors suggest that above the median score of 40, the respondent has a positive attitude towards TACs and conversely a negative attitude towards TACs for a score below 40.
To assess co-variance between oncologist and patient beliefs in TACs operating mechanisms | Inclusion
  CHBQ questionnaire completed by the oncologist at the beginning of the study (before the start of the inclusion).
  This questionnaire is composed of 10 propositions. The total score varies between 10 (total disagreement with all the proposals) and 70 (total agreement with all the proposals). The authors suggest that above the median score of 40, the respondent has a positive attitude towards TACs and conversely a negative attitude towards TACs for a score below 40.
To assess the use of TACs | inclusion, 6 month
  If individuals have used TACs, then they are offered a simplified and adapted version of the CAMP-Q (Complementary and Alternative Medicine Practitioner Use Questionnaire) completed at inclusion and 6 months after the intervention by the patient.
  This questionnaire includes 49 questions and the objective will be to evaluate if the patient has used one or more alternative medicines (1) or no alternative medicine (0). It don't have a rating
To assess satisfaction with TACs | inclusion, 6 month
  Bilateral 6-item Likert scale (-3: very dissatisfied to +3 very satisfied) at baseline and 6 months after the procedure ONLY if at least one complementary alternative technique was checked in answer n°1 of the CAMP Q questionnaire.
  This is to have a before and after evaluation.
To assess satisfaction with oncology care. | 6 month
  Two-sided 6-item Likert scale (-3: very dissatisfied to +3 very satisfied ) at 6 months post intervention. These goals are only evaluated for patients in the AFTER group
Assess patient satisfaction with the procedure. | After intervention, 6 month
  Two-way 6-item Likert scale (-3: very dissatisfied to +3 very satisfied ) evaluated after the intervention and at 6 months. This objective is only evaluated for patients in the AFTER group
Assess patient recommendation of the intervention | After intervention, 6 month
  Two-way Likert scale with 4 items (-2 not at all agree to +2 completely agree ) evaluated after the intervention and at 6 months. This objective is only evaluated for patients in the AFTER group

CONTACTS AND LOCATIONS:
Overall Officials: NICOLAS PINSAULT, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Chu Grenoble, Grenoble
  - Pole Sante Saint Martin D'Heres, Saint-Martin-d'Hères

IPD SHARING:
Plan to Share IPD: Undecided